CLINICAL TRIAL: NCT06082674
Title: Novel Low Cost Bubble CPAP as an Alternative Non-invasive Respiratory Support Among Preterm Infants With Respiratory Distress Syndrome
Brief Title: Novel Low Cost Bubble CPAP as an Alternative Respiratory Support in Low Resource Setting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ilocos Training and Regional Medical Center (Other Government)
Responsible Party: Principal Investigator, Navid Roodaki, Dr., Ilocos Training and Regional Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITRMC-REC-2022-11
Record Dates: First submitted 2023-10-03; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Premature; Respiratory Distress Syndrome in Premature Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study Blinded the investigator and outcome assesors
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vayu CPAP Group (Experimental): The patients will be hooked to VAYu bCPAP
  Interventions: Device: Vayu bCPAP
- Mechanical Ventilator Driven CPAP (Active Comparator): Patients will be hooked to Mechanical Ventilator Driven CPAP
  Interventions: Device: Mechanical Ventilator Driven CPAP

INTERVENTIONS:
Device: Vayu bCPAP — The Vayu bCPAP uses a constant flow of dry oxygen from the source with an adjustable flow meter. Oxygen is blended by Venturi blender with ambient air to create a source of oxygen-enriched air of adjustable concentration.
  Arms: Vayu CPAP Group
Device: Mechanical Ventilator Driven CPAP — Mechanical Ventilator Driven CPAP
  Arms: Mechanical Ventilator Driven CPAP

SUMMARY:
This is a single-blind randomized controlled trial done in a Level III neonatal intensive care unit. Preterm newborns with RDS were randomized to receive oxygen therapy through bubble CPAP vs ventilator-derived CPAP. Differences in arterial blood gases, oxygen saturation, number of surfactant and CPAP failure rate between study groups were analyzed.

DETAILED DESCRIPTION:
Background and Objective: Respiratory distress syndrome (RDS) among premature infants is one of the major causes of neonatal death. The use of continuous positive airway pressure (CPAP) has become a standard of care for preterm newborns with RDS. In countries faced with the challenge of improving neonatal care, cost-effective innovations for respiratory support are a promising intervention. This study determined the efficacy of a low-cost bubble CPAP as an alternative non-invasive oxygen therapy for newborn infants with RDS.

METHODS: This is a single-blind randomized controlled trial done in a Level III neonatal intensive care unit. Preterm newborns with RDS were randomized to receive oxygen therapy through bubble CPAP vs ventilator-derived CPAP. Differences in arterial blood gases, oxygen saturation, number of surfactant and CPAP failure rate between study groups were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Included are preterm neonates less than 36 weeks (WHO definition)
* admitted at NICU
* APGAR scores of > 7 in the 1st and 5th minute of life
* in respiratory distress at birth,
* radiologic findings of RDS
* Respiratory Severity Score (RSS) or Downe's score > 4 at 10-15 minutes after hooking to CPAP
* requiring CPAP or more than 40% FiO2

Exclusion Criteria:

* Infants requiring neonatal resuscitation such as bag mask ventilation, chest compression or intubation at birth
* with comorbidities such as facial anomalies, tracheoesophageal fistulas, congenital heart disease, and other congenital anomalies which may interfere with the interface of both devices.

Ages: 5 Minutes to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Partial pressure of arterial oxygen (pa02) using Arterial Blood Gas | 8 months
  Difference in the Partial pressure of arterial oxygen (pa02) using Arterial Blood Gas
Partial pressure of carbon dioxide (pC02) using Arterial Blood Gas | 8 months
  Difference in the Partial pressure of carbon dioxide (pC02) using Arterial Blood Gas
Oxygen Saturation | 8 months
  Difference in the oxygen saturation using pulse oximeter

SECONDARY OUTCOMES:
CPAP Failure | 8 months
  Difference in the number of CPAP failure
surfactant use | 8 months
  total number of surfactant use

CONTACTS AND LOCATIONS:
Overall Officials: Navid Roodaki, MD, Principal Investigator — Ilocos Training and Regional Medical Center
Locations (1):
- Ilocos Training and Regional Medical Center, San Fernando City, La Union, Philippines

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Badin S, Roodaki N, Garcia DEC, Abila-Cariaga R, Burke TF. Evaluation of a novel reprocessed bCPAP system on sepsis rates among preterm neonates with respiratory distress: a randomized controlled trial. Front Pediatr. 2025 May 19;13:1569437. doi: 10.3389/fped.2025.1569437. eCollection 2025. PMID 40458453